CLINICAL TRIAL: NCT04718519
Title: Responses of International Migrant Workers to Large-Scale Dormitory Outbreaks of COVID-19: A Population Survey
Brief Title: Migrant Workers' Responses to the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Other Study IDs: 510d2
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Coronavirus; Trust; Misinformation
Keywords: Migrant workers; Singapore; Vulnerable; Trust; Rumours; Resilience
MeSH Terms: conditions — Coronavirus Infections; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Migrant Workers

SUMMARY:
Rumors circulate widely during public health crises and have deleterious consequences. In this study, we seek to document the base rates of migrant workers' rumor exposure and identify predictors of rumor hearing, sharing and belief.

DETAILED DESCRIPTION:
Rumors circulate widely during public health crises and have deleterious consequences. Vulnerable populations such as migrant workers tend to lack access to accurate health information, which can put them at higher risk for receiving and spreading misinformation.

In this study, we seek to document (i) the base rates of migrant workers' rumor exposure and (ii) identify predictors of rumor hearing, sharing and belief. These predictors include trust in institutions, risk perceptions, online habits and socio-demographic variables.

Data was taken from the COVID-19 Migrant Health Study, a cross-sectional study of male migrants employed in manual labor jobs within Singapore.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old
* Holds a government work permit identifying their employment status

Exclusion Criteria:

* NIL

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consist of male migrant workers employed in manual labor jobs within Singapore
Sampling Method: Non-Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-10-11 (Actual); Study Completion 2020-10-11 (Actual)

PRIMARY OUTCOMES:
Confidence in government | baseline
  Participants were asked how confident they were that the government could control the nationwide spread of COVID-19
Fear for health | baseline
  Participants were asked how fearful they were about their health during the COVID-19 situation
Fear for job | baseline
  Participants were asked how fearful they were about their job during the COVID-19 situation
Degree of exposure to rumours | baseline
  We investigated participants' familiarity with five rumors that had been widely spread during the COVID-19 pandemic: (1) drinking water frequently will help prevent infection (COVID-19 prevention); (2) eating garlic can help prevent infection (COVID-19 prevention); (3) the outbreak arose from people eating bat soup (COVID-19 origins); (4) the virus was created in a US lab to affect China's economy (COVID-19 origins); and (5) the virus was created in a Chinese lab as a bioweapon (COVID-19 origins).
Online habits | baseline
  We investigated the number of hours per day that participants' spent checking COVID-19 news and discussing COVID-19 on social media.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale NUS, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Due to stipulations by the Institutional Review Board, data cannot be shared.